CLINICAL TRIAL: NCT05543967
Title: A Cross-sectional and Longitudinal Study to Establish Diagnostic Models Based on Olfactory Function and Odor-induced Brain Activation for Diabetes-Related Cognitive Impairment
Brief Title: Establish Diagnostic Models Based on Olfactory Function and Odor-induced Brain Activation for Diabetes-Related Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-PY-15
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes Mellitus; Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes Mellitus: These patients must have a definite diagnosis of type 2 diabetes mellitus (T2DM) according to the American Diabetes Association (ADA) standards. Some of these patients have symptoms of cognitive impairment, while others have normal cognition. All T2DM patients will undergo physical exam, cognitive and olfactory test as well as structural and brain functional MRI at baseline and follow-up time points.
  Interventions: Behavioral: Cognitive assessments; Other: Olfactory function measurements; Other: Functional magnetic resonance imaging
- Healthy Control: These participants have normal glucose tolerance and normal cognition. All HC subjects will undergo physical exam, cognitive and olfactory test as well as structural and brain functional MRI at baseline and follow-up time points.
  Interventions: Behavioral: Cognitive assessments; Other: Olfactory function measurements; Other: Functional magnetic resonance imaging

INTERVENTIONS:
Behavioral: Cognitive assessments — Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Rey Auditory Verbal Learning Test (RAVLT), Boston Naming Test (BNT), Digit Span Test (DST), Trail Making Test (TMT).
Other: Olfactory function measurements — Olfactory Threshold, Odor Identification Score, Odor Memory Score.
Other: Functional magnetic resonance imaging — resting-state fMRI, odor-induced fMRI.
  Other Names: fMRI

SUMMARY:
This is a cross-sectional and longitudinal study to establish diagnostic models based on olfactory function assessments and odor-induced brain activation for cognitive impairment in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Patients with diabetes have increased risks of cognitive impairment and dementia, which affecting the quality of life and diabetes management. Therefore, it is an urgent challenge to identify non-invasive biomarkers for early diagnosis and prognosis of the cognitive decline in patients with diabetes. Previous research has shown that both olfactory dysfunction and decreased odor-induced brain activation are present before clinically measurable cognitive decrements in type 2 diabetes. This is a cross-sectional and longitudinal study to establish diagnostic models based on olfactory function assessments and odor-induced brain activation for cognitive impairment in patients with type 2 diabetes mellitus. The investigators will recruit 200 patients with type 2 diabetes in the outpatient and inpatient departments. Health controls will be recruited from the community. At the baseline, clinical information collection, 100g-steamed bread meal test, biochemical measurement, cognitive assessments, olfactory test and functional magnetic resonance imaging(fMRI) scan will be conducted for all participants. Study duration was 3 years with a follow-up every 18 months. In the longitudinal study, all of the assessments will be repeated to evaluate changes of observational parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-75 years
* Right handedness
* Possessed over 6-year education
* Provision of informed consent prior to any study specific procedures
* Disease duration of T2DM patients >1 year

Exclusion Criteria:

* Control participants would be excluded if they had a fasting blood glucose level >7.0 mmol/L; glucose level> 7.8 mmol/L after oral glucose tolerance test (OGTT); HbA1c>5.7%
* Control participants would be excluded if they had a Montreal Cognitive Assessment (MoCA, Beijing edition) score of < 26
* Any acute disease
* History of neurologic or psychological illness
* Abnormal results of thyroid hormones, vitamin B12, and folate
* Metal implants, unable to complete the MR scanning
* Partial or complete olfactory dysfunction associated with sinusitis, allergic rhinitis, and deviated nasal septum
* Pregnant or lactating women
* Participating in other clinical trials at the same time or within 6 months prior to the start of the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM patients will be recruited from the outpatient and inpatient units of the endocrinology department of the investigator's hospital. Healthy control will be recruited in the community.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-18 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Baseline cognitive performance | Day 1 of entry study
  The Montreal Cognitive Assessment (MoCA) score, ranges from 0 to 30, and higher scores mean better cognition.
Baseline olfactory threshold | Day 1 of entry study
  Olfactory threshold test: score range 1-13.5, which is determined based on a series of binary dilutions of the N-butanol solution in light mineral oil. The higher the score is, the more sensitive the participant is in detecting an odor. Scores of 8-10 were considered normal olfactory sensitivity, whereas scores of 1-3 signified olfactory dysfunction or anosmia, and scores of ≥10 indicate better olfactory sensitivity.
Baseline olfactory memory | Day 1 of entry study
  Olfactory memory test: Part A: Participants are shown 4 pictures for each odor (10 odors in total), then they need to select what they sniffed. Have a 10-minute break. Part B: Participants sniff 20 different odors, 10 of which are the same odors as in Part A. They need to select the picture and figure out whether the odor is old or new.
Baseline odor-induced brain fMRI activation | Within 1 week after cognitive assessments
  Each participant underwent a series of task fMRI scans to measure temporal brain response to four increasing concentrations of lavender odors (0.032%, 0.10%, 0.32%, and 1.0) diluted in 1,2-propanediol (Sigma-Aldrich, St. Louis, MO). The visual cues of "+" and "smell" were used for baseline and odor stimulation, respectively. Each concentration was assessed three times, with fresh air and scent occurring alternately. Participants were instructed to press a button once they smelled the lavender scent. A general linear model was used to estimate odor-induced brain activation. Contrasts between "fresh air > rest" and "scent > rest" for each participant were made to get odor-induced brain activation value. Bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, entorhinal cortex, and hippocampus were extracted and merged as olfactory regions of interest (ROIs) for further analyses.
Longitudinal changes of cognitive performance | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of MoCA score from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up). The Montreal Cognitive Assessment (MoCA) score, ranges from 0 to 30, and higher scores mean better cognition.
Longitudinal changes of olfactory threshold | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of olfactory threshold tests score from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up). Olfactory threshold test: score range 1-13.5, which is determined based on a series of binary dilutions of the N-butanol solution in light mineral oil. The higher the score is, the more sensitive the participant is in detecting an odor. Scores of 8-10 were considered normal olfactory sensitivity, whereas scores of 1-3 signified olfactory dysfunction or anosmia, and scores of ≥10 indicate better olfactory sensitivity.
Longitudinal changes of olfactory memory | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of olfactory memory tests score from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up). Olfactory memory test: Part A: Participants are shown 4 pictures for each odor (10 odors in total), then they need to select what they sniffed. Have a 10-minute break. Part B: Participants sniff 20 different odors, 10 of which are the same odors as in Part A. They need to select the picture and figure out whether the odor is old or new.
Longitudinal changes of odor-induced brain fMRI activation | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of odor-induced brain activation beta value from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up)

SECONDARY OUTCOMES:
Baseline brain structural MRI scan | Within 1 week after cognitive assessments
  Cortical morphology
Baseline brain functional MRI scan | Within 1 week after cognitive assessments
  Large-scale network functional connectivity
Longitudinal changes of brain structural MRI scan | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of cortical morphology from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up)
Longitudinal changes of functional MRI scan | From baseline to 18 months' follow-up and 36 months' follow-up
  Compare the change of large-scale network functional connectivity from baseline to each follow-up time points (18 months' follow-up, 36 months' follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be made during the 12 months after the end of study, and the original data can be obtained from the PI if necessary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: during the 12 months after the end of study